CLINICAL TRIAL: NCT05104840
Title: Randomized Study on Determine the Expression of the Furin Protein in Patients With Confirmed COVID-19 Disease (in Various Phases of the Disease), Recovered From SARS-CoV-2 and Vaccinated Against Coronavirus (All Types of Vaccines)
Brief Title: A Randomized Study to Determine the Expression of the Furin Protein in Patients With SARS-CoV-2 and Vaccinated Against Coronavirus
Status: Terminated | Type: Observational
Why Stopped: the company is liquidated
Sponsor: Center Trials & Treatment (Other)
Collaborators: Oleg Martynenko (Unknown)
Responsible Party: Sponsor
Other Study IDs: 6564N20-20
Record Dates: First submitted 2021-10-28; First posted 2021-11-03 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; SARS-CoV-2; Furin; RGMc Processing; Paired Basic Amino Acid Cleaving Enzyme (PACE)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The rapid spread of SARS-CoV-2 (also known as 2019-nCoV and HCoV-19 1), a novel beta coronavirus B lineage (βCoV), has sparked a global coronavirus disease (COVID-19) pandemic. It has been suggested that RRAR, a unique furin-like cleavage site (FCS) in the spike protein (S) that is absent in other B βCoV lines such as SARS-CoV, is responsible for its high infectivity and transmissibility.

Furin is a protein with a special function of a fermentative biocatalyst: which recognizes the degree of maturity of a group of amino acids Functionally, Furin works to renew the body, but it is also a path to the introduction of the SARS-CoV virus into a living human cell, HIV virus, Ebola virus, and others that penetrate a human cell using the Furin protein, sending a conditioned signal from the extracellular matrix, and gives the virus the opportunity to merge the protein of the coronavirus spike and the protein content of the cut cell, which activates the phase of virus replication in the body.

We hypothesize that measuring the quantitative indicators of Furin protein expression in patients (at the onset of the disease) who have recovered from SARS-CoV-2 and vaccinated (with all types of vaccines) against coronavirus can provide an understanding of the molecular-cellular mechanisms of the virus's cellular invasion. This means that it will be possible to find new ways to prevent the fusion of the membranes of infected cells with normal ones (this mechanism allows the virus to spread throughout the body without leaving the affected cells).

Protein identification will be carried out by Enhanced Chemiluminescence (ECL) (the method of enhanced chemiluminescence differs from the method of immunochemical staining using chromogenic substrates by a much greater sensitivity)

DETAILED DESCRIPTION:
The parameters of the Furin protein in the blood of patients with a confirmed diagnosis of COVID-19 on days 4, 8, or 14 after the onset of symptoms of the disease or a positive PCR test will be assessed ( provided they are in a hospital or clinic for inpatient or outpatient treatment).

* Patients will be asked to donate blood for an enzyme-linked immunosorbent assay of levels of specific IgM and IgG to SARS-CoV-2 from the 3rd to the 39th day after the development of COVID-19 (provided they are in a hospital or clinic for inpatient or outpatient treatment)
* Patients will be asked to take a blood test to quantify antibodies (IgG, IgM) to the IgG class coronavirus to the SARS-CoV-2 spike (S) protein and IgM antibodies, to proteins (nucleocapsid (N) and RBD site of the S-protein ) SARS-CoV-2, (ELISA),

The presence of specific antibodies in the blood serum allows you to determine whether the body has met with the COVID-19 virus and whether antibodies have been developed during the contact that recognizes] this virus when they meet again. ⠀ The primary immune response to antigens new to the body begins with the production of immunoglobulins M (IgM). IgM to COVID-19 appears in the blood about 2-3 weeks after exposure to the virus in the case of asymptomatic COVID-19 and disappears by about 14-16 weeks.

Since the formation of antibodies is due to the individual characteristics of the immune system, the results of selective testing on different test systems in different countries in different ethnic groups should verify the result.

* The absence of antibodies will not be evidence of the absence of infection, since there is a concept of a "serological window", when the pathogen has already entered the body, the pathological process develops, but antibodies have not yet appeared.

Age data will be taken into account This study does not imply the receipt, storage and processing of personal data.

* In the vaccinated, the level of Furin protein in the blood will be determined after the first and (or) after the second vaccination, as well as after the booster dose on days 10-60-120-240-360 after vaccination.
* In those who have been ill, but not vaccinated with any vaccine against coronavirus, the level of Furin protein in the blood will be determined up to 60 days after receiving a negative PCR test and the absence of clinical signs of the disease.
* In patients with post-COVID conditions (syndrome), or with a severe form of the disease, the indicators will be determined up to day 180 inclusive after receiving a negative PCR test and the absence of acute clinical signs of the disease.
* If the patients have data, the results of genotyping / mutation and coronavirus variant will be taken into account.
* Patients may be offered compensation (financial reward) for taking tests, participating in a survey, and providing data and/or travel expenses for testing.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Age > 18
* Hospitalized adult male and female patients with Laboratory-confirmed novel coronavirus (SARS-CoV-2) infection
* Laboratory-confirmed novel coronavirus (SARS-CoV-2) infection
* All Confirmed COVID-19 Patients by PCR or highly suspected patients admitted to the chest department's isolation unit during the duration of the study
* Able to understand and provide voluntary informed consent. Informed consent for participation in the study (consent can be oral if written consent cannot be expressed
* Vaccination with any type of SARS-CoV-2 vaccine

Exclusion Criteria:

* Other medical condition other than COVID-19 or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study
* Suspected or known active systemic bacterial, viral (except SARS-CoV2 infection) or fungal infections
* Active herpes zoster infection
* Any physical examination findings and/or history of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk to the patient by their participation in the study
* Participation in other clinical trials of investigational treatments for COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients of coronavirus departments of hospitals and clinics of any specialization.
  * Hospital patients for COVID-19 treatment.
  * Patients with confirmed SARS-CoV-2 and on outpatient treatment.
  * Patients with confirmed SARS-CoV-2 and being treated at home under the remote supervision of a physician.
Sampling Method: Probability Sample
Enrollment: 2432 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Determination of the level of Furin protein in the blood of patients with confirmed SARS-CoV2 and being treated in a hospital | up to 12 month
  Determination of the level of Furin protein in the blood of patients with confirmed SARS-CoV2 and being treated in a hospital
Determination of the level of Furin protein in the blood of patients with confirmed SARS-CoV2 and who are on outpatient treatment | up to 12 month
  Determination of the level of Furin protein in the blood of patients with confirmed SARS-CoV2 and who are on outpatient treatment
Determination of the level of furin protein in the blood of those vaccinated against SARS-CoV2 after the first and second vaccinations (or after the ones-dose vaccine J&J) | up to 12 month
  Determination of the level of furin protein in the blood of those vaccinated against SARS-CoV2 after the first and second vaccinations (or after the ones-dose vaccine J&J)

SECONDARY OUTCOMES:
determination of the levels of antibodies (IgG, IgM) to the proteins (nucleocapsid (N) and the RBD S-protein site) SARS-CoV-2 in patients with test positive for COVID-19 | up to 12 month
  determination of the levels of antibodies (IgG, IgM) to the IgG class coronavirus, to the spike protein (S) SARS-CoV-2 and IgM antibodies, to the proteins (nucleocapsid (N) and the RBD S-protein site) SARS-CoV-2 in patients with test positive for COVID-19
determination of the levels of antibodies (IgG, IgM) to the proteins (nucleocapsid (N) and the RBD S-protein site) SARS-CoV-2 in vaccinated against coronavirus disease (randomized sample by type of vaccine) | up to 12 month
  determination of the levels of antibodies (IgG, IgM) to the IgG class coronavirus, to the spike protein (S) SARS-CoV-2 and IgM antibodies, to the proteins (nucleocapsid (N) and the RBD S-protein site) SARS-CoV-2 in vaccinated against coronavirus disease (randomized sample by type of vaccine)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (4):
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - StatMed Ocala, Ocala, Florida
  - Medical University of South Carolina, Charleston, South Carolina
  - Seattle Intstitute of East Asian Medicine, Seattle, Washington
- India (4):
  - Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi
  - Humsafar Trust, Mumbai
  - Max Super Speciality Hospital Saket, New Delhi
  - Sher i Kashmir Institute of Medical Sciences, Srinagar
- State Institution Republican Clinical Hospital, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after the end of the research

REFERENCES:
- See also: The role of furin cleavage site in SARS-CoV-2 spike protein-mediated membrane fusion in the presence or absence of trypsin — https://www.nature.com/articles/s41392-020-0184-0
- See also: The origin of SARS-CoV-2 furin cleavage site remains a mystery — https://www.news-medical.net/news/20210217/The-origin-of-SARS-CoV-2-furin-cleavage-site-remains-a-mystery.aspx